CLINICAL TRIAL: NCT07172334
Title: What is the Role of the Exposome in Pulmonary Hypertension
Acronym: EXPOSPAH
Status: Not yet recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A00986-43
Record Dates: First submitted 2025-09-03; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension (PAH); Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Keywords: Pulmonary hypertension; Exposome
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Surveys and Questionnaires; Sampling Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Two strands of hair (or beard or axillary hair) will be taken, along with a urine and blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAH group (cases): Patients with PAH without associated pathology: idiopathic or heritable, or with features of venous/capillary involvement, according to the clinical classification of PH
  Interventions: Other: Questionnaires; Other: Samples
- CTEPH group (controls): Patients with chronic thromboembolic PH (CTEPH, class 4), according to the clinical classification of PH
  Interventions: Other: Questionnaires; Other: Samples

INTERVENTIONS:
Other: Questionnaires — Patients will complete questionnaires on professional exposures with the help of a trained professional (estimated time: 30 minutes), followed by self-questionnaires on indoor and outdoor pollution, medications, drugs and socio-economic variables (estimated time: 30 minutes).
Other: Samples — Two strands of hair (or beard or axillary hair) will be taken, along with a urine and blood sample.

SUMMARY:
Pulmonary arterial hypertension (PAH) is a rare and incurable disease affecting people of all ages. It is characterized by obstructive remodeling of the small pulmonary arteries, responsible for an increase in pulmonary arterial pressure, leading to right heart failure and death in the absence of treatment. PAH can be associated with a variety of diseases, but around half of all PAH cases are idiopathic or hereditary, and may develop on predisposed terrain following a "second hit", as suggested by the identification of PAH cases associated with the use of anorectic drugs, methamphetamine and occupational exposure to organic solvents. No study has systematically analyzed the exposome of patients with PAH, combining environmental and occupational exposures as well as drugs and medications.

The exposome of patients with PAH without associated causes will be compared with that of patients with another form of pulmonary hypertension (PH), linked to thromboembolic risk factors: chronic thromboembolic PH (CTEPH), which will constitute the control group.

ELIGIBILITY:
Inclusion Criteria:

* Consent signed by the participant
* Age ≥ 18 years
* Free subject, under no legal protection
* Good understanding of the French language, allowing to answer the questionnaires
* Incident patients with pre-capillary PH confirmed by cardiac catheterization (PAPm > 20mmHg, PCP ≤ 15 mmHg, RVP > 2UW) having had the right diagnostic cardiac catheterization within one year (≤1 year) :

  * Cases: Patients with PAH without associated pathology: idiopathic or heritable, or with features of venous/capillary involvement, according to the clinical classification of PH
  * Controls: Patients with chronic thromboembolic PH (CTE-PTH, class 4), according to the clinical classification of PH.

Exclusion Criteria:

* Patients classified as HTP groups 2, 3 or 5
* Patients with a diagnosis of PAH associated with a connective tissue disease, HIV, portal hypertension, congenital heart disease, bilharzia, or a drug or toxic cause considered certain according to the international classification (Aminorex, Benfluorex, Carfilzomib, Dasatinib, Dexfenfluramine, Fenfluramine, Methamphetamines, Mitomycin C, adulterated rapeseed oil)
* Patients with signs of right heart failure requiring amines and/or intensive care hospitalization at time of visit (may be included at a later visit)
* Patients refusing hair sampling or having no hair > 2 cm to allow sampling
* Patients benefiting from enhanced protection, i.e. minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social establishment, adults under legal protection, and patients in emergency situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients understanding French language with pre-capillary PH confirmed by cardiac catheterization during the year (PAH without associated pathology and CTEPH class 4)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To compare the concentration of 180 environmental toxins of interest in the hair and urine of patients with newly diagnosed PAH and CTEPH, diagnosed in one of the reference or competence centers of the French PAH network. | From enrollement to the end of study at day 1

SECONDARY OUTCOMES:
Compare broad screening of hair and urine for environmental toxicants and drugs in PAH and CTEPH patients | From enrollement to the end of study at day 1
Compare each of the 4 exposure domains (toxic agents (drugs and medications), occupational exposures, environmental exposures and socioeconomic factors) individually between PAH and CTEPH patients. | From enrollement to the end of study at day 1
Compare the exposome of PAH patients and CTEPH patients, divided into 4 domains including toxic agents using a combination of direct measurements on hair and urine and indirect measurements via questionnaires. | From enrollement to the end of study at day 1
  Compare the exposome of PAH patients and CTEPH patients, divided into 4 domains including toxic agents (drugs and medications), occupational and environmental exposures and socioeconomic factors, using a combination of direct measurements on hair and urine and indirect measurements via questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Céline ABONNEAU, Project Manager, Study Chair — Poitiers University Hospital

IPD SHARING:
Plan to Share IPD: Undecided